CLINICAL TRIAL: NCT01412502
Title: Evaluation of Post Traumatic Stress Among the Nearest Relatives of Brain-dead, Withdrawal of Life Support, and Sudden Death Patients
Brief Title: Post Traumatic Stress Among Relatives of Brain-dead, Withdrawal of Life Support, and Sudden Death Patients
Status: Terminated | Type: Observational
Why Stopped: no recruitment
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: PHRC-N/2009/CB-01; 2009-A00848-49 (Other: RCB number)
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Tissue Donors; Tissue and Organ Procurement; Brain death; Withdrawal of life support
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Brain death with organ donation: Participants in this group are the nearest relatives (or "person-of-trust") of a patient who has passed away within 3 days of admission to an intensive care unit. The cause of death includes brain death with multiple organ donation +/- tissues.
  Interventions: Other: IES-R and HDAS scores
- Limitation/cessation of active treatment: Participants in this group are the nearest relatives (or "person-of-trust") of a patient who has passed away within 3 days of admission to an intensive care unit. The cause of death includes limitation/cessation of active treatment without brain death.
  Interventions: Other: IES-R and HDAS scores
- Sudden death: Participants in this group are the nearest relatives (or "person-of-trust") of a patient who has passed away within 3 days of admission to an intensive care unit. The cause of death was sudden death of a previously healthy patient (no physical or mental limitations; MacCabe score = 0) within 3 days of admission to ICU without LATA nor brain death.
  Interventions: Other: IES-R and HDAS scores

INTERVENTIONS:
Other: IES-R and HDAS scores — The Impact of Event Scale and Hospital Depression and Anxiety Score questionnaires are administered to participants.

SUMMARY:
This study concerns the nearest relatives of patients who have passed away within 3 days of admission to an ICU due to: (1) brain death with multiple organ donation +/- tissues or (2) death via limitation and / or cessation of active treatment (LATA) without brain death or (3) sudden death of a previously healthy patient (no physical or mental limitations; MacCabe score = 0) within 3 days of admission to ICU without LATA nor brain death. Our primary objective is to determine the proportion of nearest relatives at risk for post traumatic stress disorder as defined by an Impact of Event Scale score greater than 37, and to compare this factor between the three above-mentioned groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants are the nearest relatives (or "person-of-trust") of a patient who has passed away in an intensive care unit (ICU). The cause of death must fall into 1 of the following three categories: (1) brain death with multiple organ donation +/- tissues; (2) death via limitation and / or cessation of active treatment (LATA) without brain death; (3) sudden death of a previously healthy patient (no physical or mental limitations; MacCabe score = 0) within 3 days of admission to ICU without LATA nor brain death
* The participant must be one of the following (roman numerals indicate prioritization in choice of participants, if needed): (i) designated "person-of-trust"; (ii) spouse/partner of the deceased; (iii) parent of the deceased; (iv) child of the deceased; (v) sibling of the deceased.

Exclusion Criteria:

* Patient deceased after 3 days of ICU care without LATA
* The deceased was under 18 years old
* The deceased was over 70 years old
* Refusal to participated
* Participant does not speak French
* The participant is under judicial protection, under tutorship or curatorship
* The participant is deaf or mute
* The deceased has no nearest relative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are the nearest relatives (or "person-of-trust") of a patient who has passed away in an intensive care unit (ICU) due to: (1) brain death with multiple organ donation +/- tissues or (2) death via limitation and / or cessation of active treatment (LATA) without brain death or (3) sudden death of a previously healthy patient (no physical or mental limitations; MacCabe score = 0) within 3 days of admission to ICU without LATA nor brain death
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2012-06-15 (Actual); Primary Completion 2016-06-28 (Actual); Study Completion 2016-06-28 (Actual)

PRIMARY OUTCOMES:
IES-R > 37: yes/no | 6 weeks
  Impact of Event Scale score greater than 37: yes/no

SECONDARY OUTCOMES:
IES-R | 6 weeks
  Impact of Event scale score (score varying from 0 (no risk of post traumatic stress) to 88 (highest risk of post traumatic stress)).
HDAS score | 6 weeks
  Hospital Depression and Anxiety Score (varies from 0 to 21). A score >8 indicates clinically significant anxiety/depression.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Yves Lefrant, MD PhD, Study Director — Centre Hospitalier Universitaire de Nîmes; Caroline Boutin, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (6):
- France (6):
  - Hôpital Beaujon -APHP, Clichy
  - Assistance Publique - Hopitaux de Marseille, Marseille
  - CHU Lapeyronie, Montpellier
  - Hôpital Gui De Chauliac (CHU de Montpellier), Montpellier
  - Centre Hospitalier Universitaire de Nîmes, Nîmes
  - Hôpital Kremlin Bicêtre - APHP, Paris